CLINICAL TRIAL: NCT02579369
Title: A Phase 1/2 Clinical Study to Evaluate the Safety of ALLO-ASC-DFU in the Subjects With Dystrophic Epidermolysis Bullosa
Brief Title: Study to Evaluate the Safety of ALLO-ASC-DFU in the Subjects With Dystrophic Epidermolysis Bullosa
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Anterogen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALLO-ASC-EB-101
Record Dates: First submitted 2015-10-16; First posted 2015-10-19 (Estimated); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Dystrophic Epidermolysis Bullosa
Keywords: Epidermolysis Bullosa; stem cell
MeSH Terms: conditions — Epidermolysis Bullosa Dystrophica; Epidermolysis Bullosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ALLO-ASC-DFU (Experimental)
  Interventions: Other: Allogeneic mesenchymal stem cells
- Conventional Therapy (Active Comparator)
  Interventions: Device: Polyurethene Film

INTERVENTIONS:
Other: Allogeneic mesenchymal stem cells — Dressing for Dystrophic Epidermolysis Bullosa wound.
  Other Names: ALLO-ASC-DFU
  Arms: ALLO-ASC-DFU
Device: Polyurethene Film — Dressing for Dystrophic Epidermolysis Bullosa wound.
  Arms: Conventional Therapy

SUMMARY:
This is a phase I/II open-label study to evaluate the efficacy and safety of ALLO-ASC-DFU in patients with Dystrophic Epidermolysis Bullosa.

DETAILED DESCRIPTION:
ALLO-ASC-DFU is a hydrogel sheet containing allogenic adipose-derived mesenchymal stem cells. Adipose-derived stem cells have anti-inflammatory effect and release growth factors such as vascular endothelial growth factor (VEGF) and hepatocyte growth factor (HGF), which can enhance wound healing and regeneration of new tissue, finally may provide an new option in treating a Dystrophic Epidermolysis Bullosa.

ELIGIBILITY:
Inclusion Criteria:

1. Age : 10~60
2. Diagnosed with Dystrophic Epidermolysis Bullosa based on immunofluorescence test.
3. Bullous skin lesion sized over 10 cm^2
4. Test negative for Serum β-HCG pregnancy test on screening, if the subject is fertile
5. A subject who is willing to follow the protocol and provide a informed consent on screening, given that the information with respect to the clinical trial is provided.

Exclusion Criteria:

1. A subject with history of epidermoid carcinoma within a year from screening.
2. A subject who requires antibiotics due to bacterial infection on skin.
3. A subject who was dosed with oral steroid, over 0.5mg/kg a day for subjects under 18, or over 20mg in 2 weeks for subjects over 18, within 30 days prior to screening.
4. A subject treated with radiotherapy or immunosuppressants, within 30 days prior to screening.
5. A subject treated with steroids locally, within 30 days prior to screening.
6. A subject with 2-times the maximum-standardized value of ALT, AST, ALP, bilirubin, total protein
7. A subject with 2-times the maximum-standardized value of BUN, Creatinine
8. A subject with Albumin below 2.0 g/dL.
9. A subject with Hemoglobin below 6 g/dL (anemic).
10. A subject with allergic response to bovine derived protein and fibrin glue.
11. A subject administered with biologic agents or cell therapy, within 30 days prior to screening.
12. A subject administered with stem cell treatment by IV or subcutaneously to the target wound, prior to the trial
13. A subject who enrolled into another clinical trial, within 30 days prior to screening
14. A subject with serious disease that can affect on clinical trial.
15. A pregnant or breast-feeding subject.
16. A subject with history of drug abuse within 1 year of clinical significance
17. A subject who cannot proceed according to the protocol.

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2015-12-08 (Actual); Primary Completion 2016-04-01 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Area of re-epithelization | Follow up to 8 weeks

SECONDARY OUTCOMES:
Percentage of a target wound's re-epithelialization | Every time of visit for follow up to 8 weeks
Time taken to re-epithelization | Over 8 weeks
Safety assessed by clinically measured abnormality of laboratory tests and adverse events | Over 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Su Chan Kim, PhD., Principal Investigator — Gangnam Severence Hospital
Locations (1):
- Gangnam Severence Hospital, Seoul, South Korea